CLINICAL TRIAL: NCT05899595
Title: Effects of a Personalized Physical Training to Reduce Fatigue in Chronic Fatigue Patients: a Randomized Controlled Trial.
Brief Title: Effects of a Personalized Physical Training to Reduce Fatigue
Acronym: OFF2HEALTH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Laboratoire Interuniversitaire de Biologie de la Motricité (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 23CH091; ANSM (Other: 2023-A01074-41)
Record Dates: First submitted 2023-06-02; First posted 2023-06-12 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Fatigue Syndrome, Chronic
Keywords: Fatigue; Neuromuscular function; Personalized training; Physical capacity; Fatigue status
MeSH Terms: conditions — Fatigue Syndrome, Chronic; Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Personalized training group with the fatigue status (PERSO) (Experimental): The PERSO group will perform similar exercises as the RECO group but the training load will be adapted by changing the intensity (with the same volume as RECO) depending on the fatigue scores of the week. The aerobic fatigue score will set the load for the aerobic exercises and the muscle fatigue score for the resistance exercises.
  Interventions: Other: Exercise protocol
- Traditional training group following the recommendations (RECO) (Active Comparator): The RECO group will perform aerobic and resistance exercises to reach the recommendations for patients with chronic pathologies, with a moderate intensity and an increasing volume.
  Interventions: Other: Exercise protocol

INTERVENTIONS:
Other: Exercise protocol — Patients will be randomly assigned to the PERSO or the RECO group. Each week, fatigue status of the patients will be assessed with four evaluations:
  * Subjective fatigue (Rate of Fatigue scale)
  * Heart rate variability with a holter ECG
  * Muscle pain with a visual analogue scale
  * Muscle fatigue with muscular electrical stimulations with the Myocene® The two first correspond to an aerobic fatigue score and the two latter to a muscle fatigue score.
  The RECO group will perform aerobic and resistance exercises to reach the recommendations for patients with chronic pathologies, with a moderate intensity and an increasing volume.
  The PERSO group will perform similar exercises as the RECO group but the training load will be adapted by changing the intensity (with the same volume as RECO) depending on the fatigue scores of the week. The aerobic fatigue score will set the load for the aerobic exercises and the muscle fatigue score for the resistance exercises.

SUMMARY:
Chronic fatigue (CF) is a pathological fatigue over at least 6 months, without improvement after rest or sleep. In primary care, it is the major complaint in 5 to 10% of the consultations. Physical activity is an efficient therapy to help reducing this fatigue in addition to the improvement of muscular and cardiorespiratory functions. However, it remains little exploited. Yet the studies focus mainly on precise chronic pathologies with general trainings, without considering the fatigue status and reveal a large heterogeneity. Personalizing the physical training appears to be the next step in order to improve chronic fatigue patients care.

The objective of this study will be to investigate the relevance and the effects of a personalized physical training to reduce fatigue in chronic fatigue patients.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18
* Men or women
* FACIT-F score ≤ 34
* Ability to walk during 10 minutes without stopping
* Ability to receive the Myocene® stimulation protocol
* Have given written consent
* Members or beneficiaries of a social security program

Exclusion Criteria:

* Contraindication to experimental procedures
* Important health issues that would compromise the participant security during the study
* Persistent atrial fibrillation or 2nd or 3rd degree atrioventricular block
* Currently participating in an other interventional study or having so in the past thirty days
* Patient is pregnant
* Patient is unable to give an informed consent
* Patient is deprived of liberty or under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2023-09-27 (Actual); Primary Completion 2027-11-08 (Estimated); Study Completion 2027-11-08 (Estimated)

PRIMARY OUTCOMES:
The primary outcome is the change in the FACIT-F score obtained before and after the exercise procedure. | Month 1, 4
  The FACIT-F (Functional Assessment of Chronic Illness Therapy) is a short questionnaire consisting of 13 questions which the patient answers on a scale of 0 to 4. The scores are simply added together, inverting the scale for negative sentences, to give a result out of 52 points. The lower the score, the greater the fatigue.

CONTACTS AND LOCATIONS:
Overall Officials: David HUPIN, MD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- Centre Hospitalier de Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No